CLINICAL TRIAL: NCT01423136
Title: Postop Remote ECG ST-Monitoring (PROSE 3)
Brief Title: Remote Electrocardiographic (ECG) ST-Monitoring (PROSE 3)in Post-op Patients
Acronym: PROSE 3
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Other Study IDs: 2009521-01H
Record Dates: First submitted 2011-03-28; First posted 2011-08-25 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Cardiac Complication; Postoperative Complications
Keywords: Patients undergoing non-cardiac Surgery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Routine postop care + Holter Monitoring: With sham remote ECG ST Monitoring
- Routine postop care + Holter + remote ECG monitoring
  Interventions: Device: Remote ECG monitoring Spacelab SL 1050

INTERVENTIONS:
Device: Remote ECG monitoring Spacelab SL 1050 — If ischemia noted, Sx will be notified and currently accepted treatments of myocardial ischemia will be recommended.
  Groups: Routine postop care + Holter + remote ECG monitoring

SUMMARY:
In moderate to high risk patients, cardiovascular complications after surgery account for almost 60% of death after surgery. This study will randomize 140 patients into routine postop care with Holter monitoring versus routine postop care + remote ST monitoring + Holter monitoring. The response time to electrocardiographic (ECG) ST changes as well as the total ischemia time will be studied.

DETAILED DESCRIPTION:
This proposal aims to improve the process and quality of care in the postoperative period by early detection of ischemia and prompt use of accepted therapies in order to prevent postoperative myocardial infarctions (PMI) in patients undergoing non-cardiac surgery. Specifically, it aims to validate the safety and efficacy of wireless remote real-time ECG ST-monitoring in the reduction of the incidence of PMI. It extends two pilot feasibility studies into the postoperative period using wireless remote ST-monitoring for early detection of myocardial ischemia followed by preventative strategies. It is anticipated that this research will improve postoperative care by adopting generalizable and practical strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years, undergoing non-cardiac surgery with an expected LOS ≥ 2 days, who fulfills at least one of the six criteria for increased risk:

  1. History of CAD as defined by any of the following 6 criteria i. history of angina ii. prior myocardial infarction iii. prior positive exercise stress test iv. prior documentation of cardiac ischemia on nuclear stress testing v. prior coronary artery arteriographic evidence of atherosclerotic stenosis > 50% of vessel diameter vi. ECG with pathological Q waves in two contiguous leads
  2. PVD as defined by any one of the following 3 criteria:

     i. intermittent claudication (i.e. leg pain on walking that disappears in< 10 minutes on standing) that is known or likely to be due to atherosclerotic disease ii. an ankle/arm systolic BP ratio < 0.90 in either leg at rest iii. angiographic or Doppler study demonstrating >70% stenosis
  3. History of stroke (i.e. deficit that persisted for at least 1 week after onset) thought due to atherothrombotic disease (i.e. NOT a lacunar stroke, hemorrhagic stroke, nor embolic stroke secondary to atrial fibrillation)
  4. Hospitalization for CHF within 3 years of randomization
  5. Undergoing major open vascular surgery
  6. Any 3 of the following 7 risk factors i. high risk type of surgery (eg. Open Intrathoracic, intraperitoneal, or major orthopedic surgery) ii. any history of congestive heart failure iii. diabetes and currently on oral hypoglycemic agents or insulin iv. preoperative serum creatinine >175 micromol/L v. age > 70 years vi. history of TIA (i.e. that lasted less than 24 hours) vii. urgent / emergent surgery

Exclusion Criteria:

* Planned ICU admission; atrial fibrillation; left bundle branch block (LBBB); LVH with strain; pacemaker dependency interfering with ST analysis; hemodialysis; digoxin; CABG or PCI within 5 years without any recurrence of CAD by symptoms or cardiac investigations; surgery with low physiological trespasses such as digit re-implantation, nerve repair, etc.; COPD / asthma requiring bronchodilators within the last 12 months; refusal to transfusions; adverse drug reaction (ADR) to NSAIDS, beta-blockers, Ca-channel blockers, statins, nitrates; prior enrolment in PROSE.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under-going non-cardiac Sx with moderate to high risk of postoperative cardiovascular complications
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
duration of postop myocardial ischemia | 48 hours
  To determine if the duration of postoperative myocardial ischemia during real-time wireless management of ischemic ECG ST changes is half that of standard postop care, as determined by 48-hour ambulatory ECG monitoring

CONTACTS AND LOCATIONS:
Overall Officials: H. Yang, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada